CLINICAL TRIAL: NCT01577979
Title: Adolescent Vaccination in the Medical Home: Established and Innovative Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 10-1209; U01IP000310 (NIH)
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Immunization Rate
Keywords: Vaccination; Medical Home; Adolescents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reminder/Recall Strategy (Experimental): The experimental group will consist of patients randomly selected from participating clinics. Patients from private practices and the safety net provider may be exposed to a reminder/recall strategy involving text messaging. Text messages will be used to notify parents that their child is due for an immunization or well-care visit. Parents will be able to reply with one of three response options. Patients presenting to the randomly selected experimental managed care clinics for the first HPV vaccination dose will be offered the ability to provide the clinic with their preferred contact method. The preferred method of contact will be used for the second and third HPV dose reminder/recalls.
  Interventions: Behavioral: Text Message Reminder/Recall; Behavioral: Parent Preference
- Usual Care (No Intervention): The patients in the usual care group will receive the clinic's usual care in terms of immunization and well-care reminder/recall.

INTERVENTIONS:
Behavioral: Text Message Reminder/Recall — Adolescents will be randomly selected from the participating private practices and safety net organization clinics. Parents of selected adolescents will receive a text message to alert them that their child is due for a vaccine or well-care visit. The text message will provide response instructions. The responses can be one of three options: 1) the parent will call the clinic to schedule a visit, 2) the parent would like the clinic to call them to schedule a visit, or 3) the parent would like to stop any future text message reminders. Parents who would like the clinic to call them to schedule an appointment will be contacted by their child's provider to set up a visit. Parents may receive up to 3 text message reminders, unless they chose to stop any future messages.
  Other Names: Text Messaging
  Arms: Reminder/Recall Strategy
Behavioral: Parent Preference — Parents of adolescents being seen within the managed care organization's intervention clinics will be asked about their reminder method preference at their child's 1st HPV immunization. The preference options include phone call, text message, or email. The preference for contact method will be recorded and utilized for the 2nd and 3rd dose reminders. The clinics' usual method of reminder will be used for all other parents.
  Arms: Reminder/Recall Strategy

SUMMARY:
In this project, the investigators will develop, implement, and evaluate an adolescent vaccination quality improvement program, with the program designed to encourage adolescents to visit their usual primary care provider to receive vaccinations and other recommended preventive health services. This study will be conducted in different types of primary care settings, such as public, private, and managed care clinics serving adolescent patients of diverse backgrounds, and will provide important information to help guide future public health efforts to achieve high rates of immunization in adolescents.

DETAILED DESCRIPTION:
Specific Aim 1: Within different types of primary care practices (pediatric practices in public, private, and managed care settings) serving adolescent patients of diverse socioeconomic and racial/ethnic backgrounds, to assess provider and staff attitudes regarding the desirability, feasibility, and potential sustainability of evidence-based and innovative strategies to promote adolescent vaccination in primary care practices.

Specific Aim 2: Among parents of adolescents (and/or adolescent patients) seen at primary care practices, to assess knowledge of existing national and state programs to promote vaccination, and to assess attitudes regarding, perceived barriers to, and acceptability of various practice-based strategies to promote adolescent vaccination.

Specific Aim 3: To implement and evaluate the effectiveness of a multi-faceted quality improvement program to promote adolescent vaccination within the medical home.

1. Based upon findings from Specific Aims 1 and 2, develop a quality improvement program containing two or more interventions to promote adolescent vaccination.
2. Select intervention patients to receive a multi-faceted vaccination quality improvement program and usual care patients which will continue receiving usual care.
3. Compare the following primary outcome measure between intervention and usual care patients, overall and stratified by the type of practice setting: 1)percent of adolescents who received ≥ 1 or more needed vaccines or well-care visits
4. Compare the following secondary outcome measures between intervention and usual care patients, overall and stratified by practice setting: 1) percent of adolescent patients with ≥ 1 Tdap vaccine; 2) percent of adolescent patients with ≥ 1 meningococcal (MCV4) vaccine; 3) percent of adolescent patients with ≥ 1 HPV vaccine; 4) percent of adolescent patients with ≥ 3 HPV vaccines; 5) percent of adolescent patients receiving ≥ 1 influenza vaccine during the preceding influenza season; 6) percent of adolescent patients with either a documented history of varicella disease or ≥ 2 varicella vaccines; 7) percent of adolescent patients with ≥ 2 MMR vaccines; 8) percent of adolescent patients with ≥ 3 hepatitis B vaccines; 9) percent of adolescent patients with ≥ 3 poliovirus vaccines; and 10) percent of adolescent patients with ≥ 1 missed vaccination opportunity, defined as having a patient visit to a primary care practice, being eligible for vaccination, and not receiving needed vaccines.

Specific Aim 3 (Kaiser Only): Design, implement and evaluate an HPV reminder/recall intervention based on obtaining the parents' and adolescents' preferences for reminder method and recipient at the time of the first dose of HPV.

1. Compare 2nd and 3rd dose HPV vaccination rates among adolescents age 11-17 between intervention and usual care patients.
2. Assess process measures related to feasibility and fidelity of implementation

Specific Aim 4: Evaluate the effect of a multi-faceted vaccination quality improvement program on the receipt of non-vaccination clinical preventive services recommended for adolescents.

a) Compare the following outcome measures between intervention and usual care patients, overall and stratified by the type of practice setting: 1) receipt of ≥ 1 health maintenance visits within a 12 month interval; 2) receipt of blood pressure screening; and 3) growth assessment, as documented by the measurement of weight and height and calculation of body mass index at a clinic visit.

Specific Aim 5: Assess the cost to participating practices of implementing a multi-faceted vaccination quality improvement program designed to promote adolescent vaccination.

Specific Aim 6: After conducting a multi-faceted quality improvement program to promote adolescent vaccination, to assess provider and staff attitudes about the program, in particular the perceived benefits of the program and factors which may facilitate or hamper the sustainability of the program within study practices.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-17 years old
* Active patient (visit in last 2 years) of clinics in study
* Need one or more vaccines or well-care visit

Exclusion Criteria:

* Up to date on vaccines and well-care

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34581 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percent of adolescents who received ≥ 1 or more needed vaccines or well-care visits | 6 months
  Percent of adolescents who received ANY needed vaccine or well-care visit

SECONDARY OUTCOMES:
Percent of adolescent patients with 1 or more Tdap vaccine | 6 months
Percent of adolescent patients with 1 or more meningococcal (MCV4) vaccine | 6 months
Percent of adolescent patients with 1 or more HPV vaccine | 6 months
Percent of adolescent patients with 3 or more HPV vaccines | 6 months
Percent of adolescent patients receiving 1 or more influenza vaccine during the preceding influenza season | 6 months
Percent of adolescent patients with either a documented history of varicella disease or 2 or more varicella vaccines | 6 months
Percent of adolescent patients with 2 or more MMR vaccines | 6 months
Percent of adolescent patients with 3 or more hepatitis B vaccines | 6 months
Percent of adolescent patients with 3 or more poliovirus vaccines | 6 months
Percent of adolescent patients with 1 or more missed vaccination opportunity, defined as having a patient visit to a primary care practice, being eligible for vaccination, and not receiving needed vaccines | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado Denver, The Children's Hospital of Colorado
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kempe A, O'Leary ST, Shoup JA, Stokley S, Lockhart S, Furniss A, Dickinson LM, Barnard J, Daley MF. Parental Choice of Recall Method for HPV Vaccination: A Pragmatic Trial. Pediatrics. 2016 Mar;137(3):e20152857. doi: 10.1542/peds.2015-2857. Epub 2016 Feb 26. PMID 26921286
- [Derived] O'Leary ST, Lee M, Lockhart S, Eisert S, Furniss A, Barnard J, Eblovi DE, Shmueli D, Stokley S, Dickinson LM, Kempe A. Effectiveness and Cost of Bidirectional Text Messaging for Adolescent Vaccines and Well Care. Pediatrics. 2015 Nov;136(5):e1220-7. doi: 10.1542/peds.2015-1089. Epub 2015 Oct 5. PMID 26438703